CLINICAL TRIAL: NCT05852496
Title: Vit D and Peripheral Neuropathy in Taxane Naive Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Salah Hafez Mohamed, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 357167
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Vitamin D Deficiency; Peripheral Neuropathy
MeSH Terms: conditions — Vitamin D Deficiency; Peripheral Nervous System Diseases | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplement (Active Comparator): Vitamin D supplement intake for 6 months
  Interventions: Drug: Vitamin D
- Placebo group (Placebo Comparator): Group with no vitamin D supplement treatment
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — vitamin D supplement in cancer patients which receive taxane drugs with vit D deficiency and complaining from Peripheral neuropathy.

SUMMARY:
To evaluate the efficacy of vit D supplement in cancer patients which receive taxane drugs with vit D deficiency and complaining from Peripheral neuropathy

DETAILED DESCRIPTION:
Taxanes are a class of chemotherapy agents that promote the polymerization of tubulin into highly stable, intracellular microtubules. These microtubules cause cell death by interfering with normal cell division. (1,2) The first taxane developed and tested in the field of oncology was paclitaxel.(3,4 )The introduction of paclitaxel to the armamentarium of oncologic therapy in the early 1990s had a great impact on the standard of care in lung carcinoma, breast carcinoma, ovarian carcinoma, and other solid tumors. Subsequent to this development, another taxane, docetaxel was introduced. (5,6) Unfortunately, taxane therapy is associated with side effects such as peripheral neuropathy, myelosuppression, arthralgias, myalgias, and skin reactions that may adversely affect patient-reported quality of life (QOL). Peripheral neuropathy in particular can be severe. This toxicity is cumulative across the course of therapy, can be a dose-limiting toxicity, and may lead to dose reduction or cessation of therapy. (7) Peripheral neuropathies encompass disorders of peripheral nerve cells and fibers which manifest secondary to a wide range of pathologies. These nerves include cranial nerves, spinal nerve roots & ganglia, nerve trunks & division, along with nerves of the autonomic nervous system. The most frequently encountered symptoms of peripheral neuropathy include numbness and paresthesias , pain, weakness, and loss of deep tendon reflexes may accompany these symptoms. (8) Vitamin D is a fat-soluble vitamin that plays an important role in calcium homeostasis and bone metabolism, vitamin-D deficiency is associated with osteoporosis, increased risk of falls and fragility fractures. Many conflicting recent studies are now showing an association between vitamin D deficiency and cancer, cardiovascular disease, diabetes, autoimmune diseases, and depression. (9) Initial supplementation for 8 weeks with Vitamin D3 either 6,000 IU daily or 50,000 IU weekly can be considered. Once the serum 25-hydroxyvitamin D level exceeds 30 ng/mL, a daily maintenance dose of 1,000 to 2,000 IU is recommended. A higher-dose initial supplementation with vitamin D3 at 10,000 IU daily may be needed in high-risk adults who are vitamin D deficient (African Americans, Hispanics, obese, taking certain medications, malabsorption syndrome). Once serum 25-hydroxyvitamin D level exceeds 30ng/mL, 3000 to 6000 IU/day maintenance dose is recommended.(10) A 2022 ASCO meeting abstract by Chen et al reported that patients with vitamin D deficiency had more paclitaxel-induced neuropathy than those with normal vitamin D blood concentrations. (11)

ELIGIBILITY:
Inclusion Criteria:

* Any cancer patient > 18 years old receive taxane treatment

Exclusion Criteria:

* Patient which receive any line of treatment cause Peripheral neuropathy before taxane.
* Chronic disease associated with neuropathy such as diabetes mellitus, Guillain-Barre syndrome and autoimmune disease.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Grades of neuropathy according to the World Health Organization rating scale | after 6 months
  Grade 0 corresponds to no symptoms of neuropathy, grade 1 corresponds to paresthesias (a tingling, tickling or prickling sensation) and/or decreased tendon reflexes, grade 2 corresponds to severe paresthesias and/or mild weakness, grade 3 corresponds to intolerable paresthesias and /or marked motor loss, Grade 4 Paralysis

SECONDARY OUTCOMES:
The Toronto Clinical Neuropathy Score (TCNS) | after 6 months
  Valid and reliable scale for use in common non-diabetic polyneuropathies. Primarily for the feet. Most of the testing is done on or near the toes. Light touch testing is done with a 10 gm monofilament on the dorsum of the large toe